CLINICAL TRIAL: NCT06566287
Title: Immediate And Delayed Implant Placement Using Socket Shield Technique And Autogenous Dentin Graft (A Randomized Clinical Trial)
Brief Title: Immediate and Delayed Implant Placement Using Socket Shield Technique and Autogenous Dentin Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0629-2/2023
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Dental Implant; Tooth Loss; Socket Shield
MeSH Terms: conditions — Tooth Loss | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Immediate implant
- Group B (Active Comparator)
  Interventions: Other: Delayed implant

INTERVENTIONS:
Other: Immediate implant — Immediate Implant with Socket Shield Group
  Arms: Group A
Other: Delayed implant — Delayed Implant with Socket preserved with socket Shield and dentin graft Group
  Arms: Group B

SUMMARY:
One of the techniques that have been proposed to reduce the amount of bone resorption in anterior maxilla is the "socket shield (SS) ". This technique includes preservation of the facial segment of a root to be extracted and immediate implant placement. A technique of socket shield with delayed implantation using autogenous dentin graft for socket preservation, as an alternative to autogenous bone grafts, has shown predictable clinical and histological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with badly destructed or non-restorable maxillary anterior teeth when the Labial cortical plate is still intact, and the thickness was found to be <2mm in CBCT.
* Patients with health status according to American Society of Anesthesiology (ASA) I and II.
* Patients who agree to participate in the study.

Exclusion Criteria:

* Patients presenting with any systemic pathology or health condition that would inhibit the osseointegration process of the implants.
* Perforated labial cortical plate seen in CBCT.
* Patients undergoing radiation therapy or history of radiation within the last two years.
* Drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Change in implant stability | Baseline and 3 months
  The stability of each implant will be measured using the Osstell device. The ISQ value will be measured immediately at the time of surgery and after three months

SECONDARY OUTCOMES:
change in thickness of the facial cortical plate | Baseline and 3 months
  patients will be subjected to CBCT scans
Change in bone density | Baseline and 3 months
  patients will be subjected to CBCT scans

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt